CLINICAL TRIAL: NCT06966076
Title: Effect of Callisthenic Training on Mobility and ADL Performance in Spastic Diplegic Cerebral Palsy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/70
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Activities of Daily Living; Postural Control; Spasticity; Mobility
Keywords: calisthenic training; postural control; conventional PT; FES-I; dynamic gait index; TUG; berg balance scale; older adults; risk of fall; functional mobility; balance; dual task training; Otago exercise program
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calisthenic training group (Experimental): CALISTHENIC TRAINING
  CALISTHENIC EXERCISES
  COMMAND AND TARGET MUSCLE GROUP
  1. LEG RAISES (LEG STRENGTH) LIE ON YOUR BACK WITH YOUR LEGS STRAIGHT. LIFT LEGS OFF THE GROUND IN FRONT. LOWER THEM BACK DOWN WITHOUT TOUCHING THE FLOOR.
     TARGETS HIP FLEXOR
  2. SIDE LEG RAISES (LEG STRENGTH) LIE ON YOUR BACK WITH YOUR LEGS STRAIGHT. LIFT LEGS OFF THE GROUND AND TAKE IT TO SIDE MAXIMALL WITHOUT TOUCHING THE FLOOR.
     TARGETS LOWER ABS AND HIP ABDUCTORS
  3. GLUTE BRIDGES ( BACK STRENGTH) LIE ON YOUR BACK WITH YOUR KNEES BENT. LIFT YOUR HIPS OFF THE GROUND, SQUEEZING YOUR GLUTES. LOWER AND REPEAT. TARGETS GLUTES AND HAMSTRINGS.
  4. QUADRUPTED POSITION:
     ASK THE PATIENT TO RIDE YOUR KNEES PLAY 'HORSY' AND SLOWLY MOVE YOUR KNEES TO AND FRO AND SIDEWAYS SO THAT TO SHIFT WEIGHT FROM SIDE TO SIDE.
  5. WALL LEG LIFTS
  6. KNEELING
  7. Vertical Lift
  8. Squats
  Interventions: Procedure: calisthenic training
- conventional physical therapy group (Experimental): CONVENTIONAL PHYSICAL THERAPY
  CONVENTIONAL PHYSICAL THERAPY Week 1 Orientation of exercises Week 2-3 UPPER LIMB (20 MINS)
  Lifting a glass of water with elbow extended Moving objects from the table to a box Combing Hairs LOWER LIMB (20 MINS) Lifting the lower extremity and lowering in o nto a footstool sit to stand Standing up with loaded trey in hand corner hamstring stretch butterfly stretch Week 4-5 UPPER LIMB (20 MINS) Grasping and releasing objects lifting a glass of water to a level of 90° shoul der flexion with an extended elbow Moving objects from the table to a box LOWER LIMB (20 MINS) Reciprocal leg flexion and extension single leg stance Kicking a ball
  Week 5-8 UPPER LIMB (20 MINS) Opening Jars Throwing Balls Same As previous weeks LOWER LIMB (20 MINS) Squatting
  Interventions: Procedure: Conventional physical therapy group

INTERVENTIONS:
Procedure: calisthenic training — COMMAND AND TARGET MUSCLE GROUP
  1. LEG RAISES (LEG STRENGTH) LIE ON YOUR BACK WITH YOUR LEGS STRAIGHT. LIFT LEGS OFF THE GROUND IN FRONT. LOWER THEM BACK DOWN WITHOUT TOUCHING THE FLOOR.
     TARGETS HIP FLEXOR
  2. SIDE LEG RAISES (LEG STRENGTH) LIE ON YOUR BACK WITH YOUR LEGS STRAIGHT. LIFT LEGS OFF THE GROUND AND TAKE IT TO SIDE MAXIMALL WITHOUT TOUCHING THE FLOOR.
     TARGETS LOWER ABS AND HIP ABDUCTORS
  3. GLUTE BRIDGES ( BACK STRENGTH) LIE ON YOUR BACK WITH YOUR KNEES BENT. LIFT YOUR HIPS OFF THE GROUND, SQUEEZING YOUR GLUTES. LOWER AND REPEAT. TARGETS GLUTES AND HAMSTRINGS.
  4. QUADRUPTED POSITION:
     ASK THE PATIENT TO RIDE YOUR KNEES PLAY 'HORSY' AND SLOWLY MOVE YOUR KNEES TO AND FRO AND SIDEWAYS SO THAT TO SHIFT WEIGHT FROM SIDE TO SIDE.
  5. WALL LEG LIFTS IN STANDING STAND WITH YOUR SIDE FACING A WALL. LIFT YOUR LEG OUT TO THE SIDE AS HIGH AS POSSIBLE.
     LOWER AND REPEAT WITH THE OTHER LEG. TARGETS HIP ABDUCTERS
  6. KNEELING
  7. VERTICLE LIFT
  8. Squats
  Arms: calisthenic training group
Procedure: Conventional physical therapy group — CONVENTIONAL PHYSICAL THERAPY CONVENTIONAL PHYSICAL THERAPY Week 1 Orientation of exercises Week 2-3 UPPER LIMB (20 MINS) Lifting a glass of water with elbow extended Moving objects from the table to a box Combing Hairs LOWER LIMB (20 MINS) Lifting the lower extremity and lowering in o nto a footstool sit to stand Standing up with loaded trey in hand corner hamstring stretch butterfly stretch Week 4-5 UPPER LIMB (20 MINS) Grasping and releasing objects lifting a glass of water to a level of 90° shoul der flexion with an extended elbow Moving objects from the table to a box LOWER LIMB (20 MINS) Reciprocal leg flexion and extension single leg stance Kicking a ball Week 5-8 UPPER LIMB (20 MINS) Opening Jars Throwing Balls Same As previous weeks LOWER LIMB (20 MINS) Squatting
  Arms: conventional physical therapy group

SUMMARY:
Almost 2 to 3 out of every 1000 children have Cerebral palsy in Pakistan.Spastic type of CP is dominant about 75%, diplegia (40%) and hemiplegic are (35.5%).Spastic diplegics have tightness of lower limb more than upper limb.Their chief complaints are reduced mobility,impaired balance and coordination and lack of postural control and stability.Calisthenic training is sort of strengthening exercises in which patient use his/her own body weight as a resistance.

Calisthenic training aims to reduce movement limitation,contracture formation and improves patient's mobility for daily transfers and ambulation,active participation of patient in indoor and outdoor activities and enhance postural stability and controle during routine tasks. The current study aims to determine the effects of calisthenic training on mobility and ADL performance in spastic diplegic cerebral palsy children aged 5-12 years fulfilling the GMFCS criteria levels 1-3. A randomized control trial will be conducted in multidisciplinary lab of FUCP, department of physical medicine and peads and rehabilitation of Fauji Foundation Hospital on the sample of 32 participants. The subjects will be randomized into two groups by sealed opaque envelope method. Baseline assessment would be done by using WEEFIM measurement assessment scale for mobility and ADL performance, pediatric balance assessment Scale for postural control. Data will be collected at baseline before intervention, after 3 weeks and finally after 6 weeks of intervention. Interventional group will be receiving calisthenic training and conventional physical therapy while control group will be receiving conventional physical therapy alone. Exercise training would be done for a total of 12 sessions for 6 weeks, twice a week with each session lasting 45 minutes. Analysis would be done by using SPSS version 21. Ethical approval will be obtained from ERC of FUSH. Informed written consent will be obtained from all participants.

DETAILED DESCRIPTION:
OBJECTIVES OF STUDY

1. To determine the affects of callisthenic exercises in comparison to conventional physical therapy on mobility, ADL perfrmance and quality of life in spastic diplegic cp children .
2. To determine the affects of callisthenic exercises in comparison to conventional physical therapy on postural controle in spastic diplegic cp

HYPOTHESIS:

Alternate hypothesis:

* affect of calisthenic training in comparison to conventional physical therapy on mobility in spastic diplegic cp patients (p<0.05).
* 2HA- There will be statistically significant difference in the affect of calisthenic training in comparison to conventional physical therapy to improve ADL performance in spastic diplegic cp patients (p<0.05).
* 3HA- There will be statistically significant difference in the effect of calisthenic training in comparison to conventional physical therapy to improve postural controle in spastic diplegic cp patients (p<0.05).

NULL HYPOTHESIS

* 1H0 -There will be no statistically significant difference in the effect of calisthenic training in comparison to conventional physical therapy to improve ADL performance in spastic diplegic cp patients (p<0.05).
* 2H0 -There will be no statistically significant difference in the effect of calisthenic training in comparison to conventional physical therapy to improve mobility in spastic diplegic cp patients (p<0.05).

  3H0 -There will be no statistically significant difference in the effect of calisthenic trainingin comparison to conventional physical therapy to improve postural controle in spastic diplegic cp patients (p<0.05).

Significanve of study:

As there is no any Conclusive evidence of calisthenic training more precisely for spastic diplegic cp children so this study will be helpful for patients and other health care proffessionals to implement this study in their clinical practice and for the patients in a way they can keep continue this treatment protocol in their home bound friendly environment by using their own body weights as a resistance after quiting from sessions of this research .

it will provide a treatment protocol for targeting calisthenic training to improve mobility, incorporate postural corrections and functional capacitance in spastic cp children .

This study will maximize the indoor functional independency in the cerebral palsy

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 13 years
* Able to accept and follow verbal instructions
* Able to participate in a training program
* Based on Gross Motor Function Classification System (GMFCS SCALE 1,2 and 3)

Exclusion Criteria:

* If they have controlled seizures
* If they suffered from any inflammatory, infectious diseases, cognitive deficiencies and any musculoskeletal deformity with chronic contracture that interfere with physical activity.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
mobility | 8 weeks
  The WeeFIM was used, it is an 18-item, 7-level ordinal scale. Each item is scored on a 7-level scale, with the total score ranging from 18 (lowest) to 126 (highest).
Activities of Daily Living Performance | 8 weeks
  Will be measured by weefim functional independence measure scale. It is an 18-item, 7-level ordinal scale.
  Each item is scored on a 7-level scale, with the total score ranging from 18 (lowest) to 126 (highest).

SECONDARY OUTCOMES:
Postural control | 8 weeks
  Will be assessed by paediatric assessment scale It has 14 items and 5 level scale.1 indicating complete dependence and 5 indicating complete independence total score are 56.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan